CLINICAL TRIAL: NCT00477334
Title: A Randomized, Multicenter, Double-blind Study to Compare the Efficacy of Single-day Treatment (1000 mg b.i.d.) With Famciclovir Compared to That of Placebo in Patient-initiated Episodic Treatment of Recurrent Genital Herpes in Immunocompetent Black Patients
Brief Title: Patient-initiated Episodic Treatment of Recurrent Genital Herpes in Black Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFAM810A2310
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Genital Herpes
Keywords: Recurrent genital herpes; Black population
MeSH Terms: conditions — Herpes Genitalis | interventions — Famciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Famciclovir 1000 mg; twice a day for one day.
  Interventions: Drug: Famciclovir
- 2 (Placebo Comparator): Placebo; twice a day for one day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famciclovir — oral; two 500 mg tablets twice a day; single day treatment
  Other Names: Famvir
  Arms: 1
Drug: Placebo — oral; two tablets twice a day; single day treatment
  Arms: 2

SUMMARY:
This study will evaluate the safety and efficacy of single-day famciclovir episodic treatment in Black patients with recurrent genital herpes

ELIGIBILITY:
Inclusion Criteria:

* Black men or women 18 years or older
* History of recurrent genital herpes with at least 4 recurrences in preceding 12 months or in preceding 12 months prior to using suppressive antiviral therapy
* Documented herpes simplex virus type 2 (HSV-2) seropositivity
* Willingness to discontinue suppressive therapy during study, if applicable
* Willingness and ability to comply with the study protocol

Exclusion Criteria:

* Pregnant or breastfeeding women
* Women of childbearing potential not using accepted methods of contraception
* Hypersensitivity to famciclovir or drugs with similar chemical structures
* Renal dysfunction
* Known or suspected to have decompensated liver disease
* Known to have gastrointestinal malabsorption
* Known to be immunocompromised
* Known to be hypersensitive to ingredients in study medication
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalu Mohammed, Dr, Principal Investigator — Clayton Research Institute
Locations (43):
- United States (33):
  - Providence Clinical Research, Burbank, California
  - Alia Clinical Research, INC, Huntington Park, California
  - Dermatology Research Associates, Los Angeles, California
  - The Conant Foundation Quest Diagnostics, San Francisco, California
  - Medical Research Centers of South Florida, Inc., Hollywood, Florida
  - First Coast Primary Care Minority Physicians Research Alliance, Jacksonville, Florida
  - AppleMed Research Inc., Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Segal Institute for Clinical Research Heathcare Clinical Data, Inc, North Miami, Florida
  - Perimeter Institute for Clinical Research Inc. ("PICR"), Atlanta, Georgia
  - Medical College of Georgia Hospital and Clinics, Augusta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Clinical Trials Management LLC, Covington, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Omni Fertility and Laser Institute, Shreveport, Louisiana
  - International Research Center, Towson, Maryland
  - Miray Medical Center, Brockton, Massachusetts
  - Pearl Medical Group, PLLC, Southfield, Michigan
  - Dr. Mohammed, St Louis, Missouri
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - Metrolina Internal Medicine Internal Medicine Research, Charlotte, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - UNC Clinical Research, Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Planned Parenthood of Arkansas and Eastern Oklahoma, Tulsa, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Women's Care Center, PLC: Research Memphis Associates, Memphis, Tennessee
  - Private Practice, Fort Worth, Texas
  - R/D Clinical Research, Inc, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Millennium Clinical Trials, LLC, Arlington, Virginia
- South Africa (10):
  - Josha Research, Bloemfontein
  - Prime Cure Medicentre, Durban
  - Umkomaas Clinical Research Site, eMkhomazi
  - Drs. Essack and Mitha, Johannesburg
  - Medunsa Clinical Research Unit (MeCRU), Medunsa
  - Bertoni Mercy Clinic, Mmakau Village GA Rankuwa
  - Global Clinical Trials, Port Elizabeth
  - Eastmed Clinical Trial Centre/Eastmed Medical Centre, Pretoria
  - Setshaba Research Centre, Shoshanguve
  - Drs. AE and QE Bhorat, Soweto

REFERENCES:
- [Derived] Leone P, Abudalu M, Mitha E, Gani M, Zhou W, Hamed K. One-day famciclovir vs. placebo in patient-initiated episodic treatment of recurrent genital herpes in immunocompetent Black patients. Curr Med Res Opin. 2010 Mar;26(3):653-61. doi: 10.1185/03007990903554471. PMID 20070143
- See also: Click here for more information on this study — http://www.novartisclinicaltrials.com/webapp/etrials/DiseaseID58/Genital-Herpes-clinical-trials.go

RESULTS

PARTICIPANT FLOW:
Groups:
- Famciclovir 1000 mg: Famciclovir 1000 mg; twice a day for one day for treatment.
- Placebo Comparator: Placebo twice a day for one day for treatment.
Period: Overall Study
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Started | 312 | 151
Randomized and Took Study Drug | 206 | 98
Intent to Treat Population | 201 | 98
Participants Completing First Recurrence | 187 | 92
Modified Intent to Treat Population | 152 | 78
Completed | 142 (Participants completing the first recurrence and follow-up.) | 75 (Participants completing the first recurrence and follow-up.)
Not Completed | 170 | 76
Not completed — Discontinued prior to taking study drug | 106 | 53
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 15 | 4
Not completed — Administrative Problems | 39 | 15
Not completed — Protocol Violation | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Famciclovir 1000 mg | Placebo Comparator | Total
Number analyzed (Participants) | 201 | 98 | 299
Age Continuous [Mean (Standard Deviation); unit: years] — Intent to Treat population consists of all randomized participants who initiated treatment with the study drug with the intention of treating genital herpes recurrences
  years | 37.5 (10.35) | 38.5 (10.34) | 37.8 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent to Treat population consists of all randomized patients who initiated treatment with the study drug with the intention of treating genital herpes recurrences
  Participants
    Female | 127 | 69 | 196
    Male | 74 | 29 | 103
Number of Years: recurrent genital herpes [Mean (Standard Deviation); unit: Years] — Number of years the participant has experienced recurrent genital herpes. Intent to Treat population consists of all randomized participants who initiated treatment with the study drug with the intention of treating genital herpes recurrences
  Years | 6.9 (6.75) | 7.0 (6.50) | 7.0 (6.66)
Genital herpes recurrence in last 12 months [Mean (Standard Deviation); unit: Genital herpes recurrences] — Number of genital herpes recurrences during the last 12 months or in the 12 months immediately preceding suppressive treatment.
  Intent to Treat population consists of all randomized participants who initiated treatment with the study drug with the intention of treating genital herpes recurrences
  Genital herpes recurrences | 6.0 (3.26) | 5.8 (2.72) | 5.9 (3.09)

OUTCOME MEASURES:

1. Primary Outcome: Investigator Assessed Time to Healing of All Non-aborted Genital Herpes Lesions
Description: Time to healing of all non-aborted genital herpes lesions, defined as the time from the first dose of study medication to the investigator-assessed time of healing (i.e. loss of all crusts and re-epithelialization of lesions; erythema may be present).
Time Frame: 21 days
Population: Modified Intent to Treat Population (mITT) that includes all Intent to Treat participants with non-aborted genital herpes lesions during the treatment period.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Number analyzed (Participants) | 152 | 78
Days | 5.38 [3.82 to 7.35] | 4.79 [3.56 to 7.03]
Statistical Analysis 1: Comparison: Famciclovir 1000 mg vs Placebo Comparator; Participants who discontinued from the study before healing of non-aborted lesions was confirmed and participants who completed the study 21 days since treatment initiation without non-aborted lesion stages and without a final assessment on aborted lesion status are imputed according to the distribution of the time to healing among the subjects in the placebo group whose time to healing is greater than or equal to the observed discontinuation time. (Censor time); Test type: Superiority or Other; p = 0.4161, Hodges-Lehman Shift Model; Median Difference (Final Values) = 0.26, 95% CI 2-sided [-0.40 to 0.98] — Difference in time to healing= time to healing for Famciclovir-time to healing for Placebo. Hodges-Lehman shift model is used to estimate the difference in treatment effect. P-value is from the Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Famciclovir 1000 mg vs Placebo Comparator; Participants who discontinued from the study before healing of non-aborted lesions was confirmed and participants who completed the study after 21 days since treatment initiation without non-aborted lesion stages and without a final assessment on aborted lesion status were censored at the time of the last clinical lesion observation; Test type: Superiority or Other; p = 0.9372, Kaplan-Meier & Cox Regression; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.74 to 1.39] — Hazard ratio in time to healing=hazard rate of Famciclovir/hazard rate of Placebo. Based on Cox proportional hazards model with treatment, pooled center and gender as explanatory variables

2. Secondary Outcome: Percentage of Participants With Aborted and Non-aborted Genital Herpes Lesions During the Treatment Period
Time Frame: 21 days
Population: Intent-to-Treat (ITT). All randomized participants who initiated treatment (i.e. received any dose of the study drug) with the intention of treating genital herpes recurrences.
Measure: Number; unit: Percentage of Participants
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Number analyzed (Participants) | 201 | 98
Percentage of Participants
  Percentage with aborted lesions (n=49,20) | 24.4 | 20.4
  Percentage with non-aborted lesions (n= 152,78) | 75.6 | 79.6

3. Secondary Outcome: Investigator Assessed Time to Healing of All Non-aborted and Aborted Genital Herpes Lesions
Description: Kaplan-Meier estimation.
Time Frame: 21 days
Population: ITT participants who discontinued from the study before healing of non aborted lesions was confirmed and participants who completed the study after 21 days since treatment initiation without non aborted lesion stages and without a final assessment on aborted lesion status were assumed as having non aborted lesions in this analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Number analyzed (Participants) | 201 | 98
Days | 4.13 [1.24 to 6.00] | 4.06 [2.01 to 6.64]

4. Secondary Outcome: Time to Resolution of Symptoms Associated With Recurrent Genital Herpes
Description: Median time to resolution of symptoms: all symptoms, pain, burning, itching, tingling and tenderness associated with recurrent genital herpes estimated using Kaplan-Meier method.
Time Frame: 72 hour after initiation of study medication up to 21 days
Population: Intent to Treat Population. If a participant never had a symptom prior to the last valid diary entry for the first recurrence, then the time to resolution of the symptom was set to missing and the participant was not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Number analyzed (Participants) | 201 | 98
Days
  All symptoms (n=195/98) | 4.5 [2.8 to 8.2] | 5.7 [2.8 to 9.0]
  Pain (n=141,69) | 3.0 [1.5 to 5.3] | 2.6 [1.5 to 5.9]
  Burning (n=126,65) | 2.3 [1.0 to 4.0] | 2.5 [1.5 to 4.4]
  Itching (n=168,86) | 3.2 [1.5 to 6.0] | 3.5 [1.6 to 6.6]
  Tingling (n=141,70) | 2.0 [1.0 to 4.2] | 2.3 [1.1 to 5.9]
  Tenderness (n=147/74) | 3.4 [1.6 to 6.5] | 2.9 [1.6 to 6.0]

5. Secondary Outcome: Number of Participants With a Second Recurrence of Genital Herpes in the Follow-up Period
Description: Number of participants with a second recurrence of genital herpes in the follow-up period.
Time Frame: 6 months
Population: Intent to Treat Population: participants who completed the first recurrence.
Measure: Number; unit: Participants
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Number analyzed (Participants) | 185 | 92
Participants | 141 | 75

6. Secondary Outcome: Time to Second Recurrence of Genital Herpes
Description: Kaplan Meier estimated time in days to second recurrent from treatment initiation and from the date of healing of aborted lesions.
Time Frame: 6 months
Population: Intent to Treat Population: participants who completed the first recurrence.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Number analyzed (Participants) | 185 | 92
Days
  Time from initiation of treatment | 69.0 [31.0 to 143.0] | 81.0 [31.0 to 122.0]
  Time from healing of non-aborted lesion | 63.0 [25.0 to 137.0] | 75.0 [24.0 to 118.0]

7. Secondary Outcome: The Number of Participants With Clinically Notable Shifts From Normal at Baseline by Hematology Test and Treatment
Description: The number of participants with clinically noted shifts in Hematology tests from normal at baseline are graded based on Division of Microbiology and Infectious Diseases (DMID) toxicity tables from Grade 1 toxicity (smallest change) to Grade 4 toxicity (largest change). Grade 3 and 4 toxicities are considered to be clinically meaningful.
Time Frame: Baseline, Day 2
Population: 304 Participants = 206 participants in the Famciclovir Group + 98 participants in the Placebo Group. Individual n values in each of the categories is the number of participants in the group with normal baseline values and at least one non-missing post baseline measurement.
Measure: Number; unit: Participants
Arm/Group | Grade 1 Toxicity | Grade 2 Toxicity | Grade 3 Toxicity | Grade 4 Toxicity
Number analyzed (Participants) | 304 | 304 | 304 | 304
Participants
  Haematocrit-Famciclovir (n=186) | 0 | 0 | 0 | 0
  Haematocrit-Placebo (n=87) | 0 | 0 | 0 | 0
  Haemoglobin-Famciclovir (n=183) | 2 | 0 | 0 | 0
  Haemoglobin-Placebo(n=88) | 3 | 0 | 0 | 0
  Absolute Neutrophils-Famciclovir (n=177) | 6 | 2 | 0 | 1
  Absolute Neutrophils-Placebo (n=83) | 0 | 0 | 1 | 0
  WBC(total)-Famciclovir (n=163) | 15 | 1 | 0 | 0
  WBC(total)-Placebo(n=98) | 6 | 1 | 0 | 0
  Platelet count-Famciclovir (n=184) | 0 | 0 | 0 | 0
  Platelet count-Placebo (n=88) | 0 | 0 | 1 | 0

8. Secondary Outcome: The Number of Participants With Clinically Notable Shifts From Normal at Baseline by Chemistry Test and Treatment
Description: The number of participants with clinically noted shifts in Clinical Chemistry tests from normal at baseline are graded based on Division of Microbiology and Infectious Diseases (DMID) toxicity tables from Grade 1 toxicity (smallest change) to Grade 4 toxicity (largest change). Grade 3 and 4 toxicities are considered to be clinically meaningful.
  SGPT(ALT)= Serum Glutamic Pyruvate Transaminase (Alanine Aminotransferase) and SGOT(AST)= Serum Glutamic Oxalacetic Transaminase (Aspartate Aminotransferase)
Time Frame: Baseline, Day 2
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Grade 1 Toxicity | Grade 2 Toxicity | Grade 3 Toxicity | Grade 4 Toxicity
Number analyzed (Participants) | 304 | 304 | 304 | 304
Participants
  SGPT(ALT)-Famciclovir (n=183) | 3 | 0 | 0 | 0
  SGPT(ALT)-Placebo (n=92) | 1 | 1 | 0 | 0
  SGOT(AST)-Famciclovir (n=190) | 4 | 1 | 0 | 0
  SGOT(AST)-Placebo (n=92) | 0 | 2 | 0 | 0
  Blood Urea Nitrogen-Famciclovir (n=196) | 0 | 0 | 0 | 0
  Blood Urea Nitrogen-Placebo (n=95) | 0 | 0 | 0 | 0
  Creatinine-Famciclovir (n=182) | 16 | 0 | 0 | 0
  Creatinine-Placebo (n=90) | 5 | 0 | 0 | 0
  Bilirubin(total)-Famciclovir (n=192) | 1 | 0 | 0 | 0
  Bilirubin(total)-Placebo (n=93) | 1 | 0 | 0 | 0
  Amylase-Famciclovir (n=152) | 6 | 2 | 0 | 0
  Amylase-Placebo (n=72) | 3 | 1 | 0 | 0
  Lipase-Famciclovir (n=190) | 2 | 3 | 1 | 0
  Lipase-Placebo (n=90) | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Description: AEs presented in this section are the AEs greater than 1% that occured in the treatment period. SAEs presented in this section are these that were reported either during the treatment or follow-up period (one SAE was reported during the follow-up period).
Arm/Group | Famciclovir 1000 mg | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 2/206 | 1/98
Other Adverse Events (participants affected / at risk) | 26/206 | 11/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir 1000 mg (N=206) | Placebo Comparator (N=98)
Heart Palpitations (Cardiac disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir 1000 mg (N=206) | Placebo Comparator (N=98)
Headache (Nervous system disorders) | 10 | 2
Nausea (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Blood Pressure increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Adnexa uteri pain (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.